CLINICAL TRIAL: NCT06422338
Title: A Multi-country, Two-arm, Open-label, Superiority, Randomised Controlled Trial to Study the Performance of a Rapid Triage Test Compared to Standard of Care (IMCI-based) to Guide Admission/Discharge Decisions During the First Clinical Assessment of Children With Fever
Brief Title: A Rapid Triage Test to Improve Risk-stratification of Febrile Children (EChiLiBRiST, Clinical Trial 1, Outpatients)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EChiLiBRiST CT1
Record Dates: First submitted 2024-05-10; First posted 2024-05-21 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Infectious Disease; Febrile Illness; Child, Only
Keywords: biomarkers; severity; point-of-care; triage; sub-Saharan Africa
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMCI-enhanced by suPAR levels (SoC + suPAR POC). (Experimental): IMCI-guidelines (standard of care) + Point-Of-Care (POC) test based on suPAR quantification
  Interventions: Other: IMCI-enhanced by suPAR levels (SoC + suPAR POC)
- IMCI alone (No Intervention): IMCI-guidelines (standard of care)

INTERVENTIONS:
Other: IMCI-enhanced by suPAR levels (SoC + suPAR POC) — IMCI-guidelines (standard of care) + Point-Of-Care (POC) based on suPAR quantification
  Arms: IMCI-enhanced by suPAR levels (SoC + suPAR POC).

SUMMARY:
The overall aim of the study is to provide evidence that introducing novel biomarkers evaluation at triaging (first clinical assessment), in combination with IMCI-based guidelines (SoC), is a viable strategy to enhance rapid and accurate identification of febrile children at increased risk of life-threatening infections compared to IMCI-based strategies alone (SoC), and to demonstrate whether this results in enhanced decisions of admission/referral vs discharge, and enhanced overall health outcome of children with acute fever in sub-Saharan Africa.

DETAILED DESCRIPTION:
This is a multi-country, open label, two-arm, parallel-group, superiority, individually randomised clinical trial involving 2,606 febrile children per country (two countries, total n=5212). The trial will compare the performance of a point-of-care rapid triage test (POC-RTT) based on suPAR levels (i.e.suPARnostic®) (in combination with IMCI-based strategies, which are the SoC) to appropriately support admission/referral vs discharge decisions during the first clinical assessment of febrile children aged 2-<60 months compared to the standard of care based on IMCI guidelines.

Febrile children meeting the study eligibility criteria will be randomly allocated (1:1) to one of the two triaging approaches (arms): 1) IMCI-based standard of care (SoC); or 2) IMCI-enhanced by suPAR levels (SoC + suPAR POC). Blood will be collected from all participants and only those randomised to the intervention arm (arm 2) will have suPAR levels determined at the POC using suPARnostic® device.

At baseline, all children will undergo two clinical assessments. Primary composite endpoint of "appropriateness of discharge" will be based on the first clinical assessment, which is more representative of real-world clinical practice. However, the ultimate decision on admission/referral vs discharge will be based on the second clinical assessment, which will ensure the safest possible clinical practice in the context of a clinical trial.

1. At baseline, during the first clinical assessment, all participants will be evaluated following the SoC based on IMCI guidelines, which will guide management decisions, including clinical diagnosis and treatment. This IMCI-guideline based evaluation during this first clinical assessment will be conducted by a health worker as per routine clinical practice in the outpatient departments of each study site.

   1. In the participants randomised to the control arm, decision of admission/referral vs discharge home will be informed by IMCI-based evaluation alone (SoC).
   2. In the participants randomised to the intervention arm, decision of admission/referral vs discharge home will be informed by IMCI-based evaluation enhanced by suPAR levels (SoC + suPAR POC). Clinicians will be instructed to admit for further observation any child with suPAR levels equal or superior to 4 ng/mL (except for confirmed malaria, that it will be equal or superior to 6 ng/mL), as these patients are at moderate or high risk of adverse outcomes and death. On the other hand, children with suPAR levels below 4 ng/mL (or below 6 ng/mL in case of confirmed malaria) will be eligible for discharge home at the criteria of the clinician, considering the signs and symptoms found, and based on IMCI guidelines. Hence, should clinicians in charge deem that any of these children still require admission, they will be instructed to continue with the admission regardless of suPAR levels.

   The study intervention will be implemented during the first clinical assessment, and consequently, primary composite endpoint of "appropriateness of discharge" will be based on the decision of admission/referral vs discharge home during this first clinical assessment, which is more representative of routine clinical practice in each study site.
2. All randomised participants will be also evaluated by an independent study physician in a second clinical assessment, for the implementation of a systematised clinical evaluation (IMCI-based) to uncover any danger signs or severity criteria potentially missed or misinterpreted during the first assessment. This second assessment will also include clinical variables of the clinical scores ED-PEWS, LqSOFA and LODS, as well as temperature and oxygen saturation measures. Hence, study clinicians during this second clinical assessment might be able to uncover more symptoms and signs that are admission criteria due to the tools available in the context of this clinical trial. Initially discharged patients from both arms showing a danger sign during this second assessment will be admitted, as well as those from the intervention arm with suPAR high-risk (red light) and moderate-risk (yellow light) levels, in case that the first clinician might not have adhered to the protocol during the first assessment. On the other hand, this second assessment will not overturn the decision of the first clinician if admission has been decided in case of low-risk (suPAR levels below 4 ng/mL; or below 6 ng/mL in case of confirmed malaria).

This second clinical assessment will guide the ultimate decision on admission/referral vs discharge in order to ensure the safest possible clinical practice in the context of a clinical trial.

Moreover, those participants with respiratory symptoms will be eligible for the respiratory tract infection (RTI) sub-study, where digital lung auscultations, a mid-turbinate nasal swab and a saliva sample will be collected.

Throughout the study, all participants will receive treatment as per the routine clinical practice and SoC for each diagnosis at each study site, administered by clinical staff routinely working in the participating facilities.

All participants will have follow-up evaluations by study clinicians on days 3 and 7 post-enrolment, or at any time in-between in case of clinical deterioration according to caregivers' evaluation. All participants will be also followed-up on day 28 for an interview to follow-up on serious adverse events (SAEs), as well as to collect information on secondary consultations and hospitalisation, or death. A follow-up extra visit at day 91 (month 3) can be conducted for an interview to ask for hospitalisation or death.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥2 months and <60 months
* Written informed consent from the child's parent or caregiver
* History of fever for ≤7 days OR hypothermia (i.e., axillary temperature <35.5ºC) OR suspected severe infection (e.g., in children with moderate or severe acute malnutrition).
* Lives within the catchment area of the study facility and must intend to continue to reside there for the duration of the study
* For the RTI sub-study only: presence of respiratory symptoms compatible with RTI.

Exclusion Criteria:

* Weight less than 2.5kg
* Main reason for consultation is an injury, trauma or acute poisoning
* Enrolled in another clinical trial testing a new drug
* Enrolled in a vaccine trial in the last 3 months.
* Any other condition determined by the investigators that makes it unlikely that the participant would complete the study

Ages: 2 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5212 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Appropriateness of discharge | Up to day 7
  The primary outcome is the proportion of "appropriateness of discharge" according to the first clinical assessment of febrile children aged 2-<60 months compared among the 2 study arms.
  Inappropriate discharge is defined as a composite of (fulfilling at least one of the following):
  1. Presence at baseline of World Health Organization (WHO)-proposed danger signs in discharged children; OR
  2. Presence of WHO-proposed danger signs on day 3 post-discharge; OR
  3. Requirement for additional visit at the health facility or admission at day 7; OR
  4. Death on day 7 post-discharge. The absence of any of these endpoints will be considered an appropriate discharge.

SECONDARY OUTCOMES:
Secondary consultations or admissions | Up to day 28
  Proportion of secondary consultations or admissions on day 7 and day 28 among the two study arms.
Mortality | Up to day 28
  Proportion of mortality on day 7 and day 28 among the two study arms.
Referrals to higher level facilities | Up to day 28
  Proportion of referrals of mild infections to higher level facilities at day 7 and day 28 among the two study arms.
Severe disease | Up to day 7
  Proportion of participants diagnosed with severe disease as described in IMCI (i.e. very severe diseases, severe pneumonia, severe dehydration, severe persistent diarrhoea, very severe febrile diseases, severe complicated measles, complicated severe acute malnutrition, mastoiditis, and severe anaemia), at day 3 and day 7 among the two study arms.
Symptoms duration | Up to day 28
  Median time to symptoms resolution among the two study arms until day 28.
Hospital stay length | Up to day 28
  Median length of hospital stay among the two study arms until day 28
Serious adverse events | Up to day 28
  Proportion of serious adverse events (SAEs) at day 3, day 7, and day 28, among the two study arms.
Discharge in the major aetiological diagnosis | Up to Day 28
  Proportion of "appropriateness of discharge decision" for the major aetiological diagnosis, including: malaria, respiratory and gastrointestinal infections, as well as in malnourished children, and HIV positive children, among the two study arms.
Biomarkers reduction of outcomes | Up to Day 28
  Proportion of "appropriateness of discharge decision" based on IMCI guidelines enhanced by suPAR levels quantified using B-Triage and other markers, compared to the clinical scores ED-PEWS, LqSOFA and LODS.
Admissions in the routine care | Up to Day 28
  Proportion of secondary consultations or admissions and mortality in the two study arms compared to available routine healthcare data.
Biomarkers in admitted | Up to Day 28
  Levels of suPAR and sTREM-1 and other circulating markers of endothelial function, angiogenesis, inflammation and intestinal barrier function at baseline and day 3 in plasma samples, and their association with admission.

OTHER OUTCOMES:
Secondary consultations or admission | Up to day 91
  Proportion of secondary consultations or admissions on day 91 (month 3) among the two study arms
Mortality | Up to day 91
  Proportion of mortality on day 91 (month 3) among the two study arms.
Sensitivity and specificity of POC | Up to day 28
  Sensitivity and Specificity of a POC test based on sTREM-1 to predict 28-day mortality and other severity outcomes in febrile children.
Endothelial activation markers in children with suspected Respiratory Tract Infections | Up to day 28
  Levels of immune and endothelial activation markers, including mucosal markers, in children with suspected Respiratory Tract Infections at baseline and day 3 in saliva samples, and their association with severity and antibiotic treatment.
Mucosal markers and species of bacteria and virus in children with Respiratory Tract Infections | Up to day 7
  Species of bacteria and virus present in the mucosa of children with Respiratory Tract Infections and their association with specific mucosal markers, susceptibility and prognosis of infection

CONTACTS AND LOCATIONS:
Overall Officials: Quique Bassat, Prof, Principal Investigator — Barcelona Institute for Global Health
Locations (1):
- Mopeia Sede Health Centre, Mopeia, Mozambique

IPD SHARING:
Plan to Share IPD: Yes
This clinical trial, as part of the wider EChiLiBRiST project, is committed to European Union-funded Horizon 2021 aims to improve and maximize access to and reuse of research data generated by the Project.
  Biological samples and data will be shared using material and data transfer agreements with the collaborating institutions.
  The full protocol will be available on request to any interested professional and may be published in peer-reviewed journals or deposited in an online repository. A fully de-identified data set of the complete patient-level data will be available for sharing purposes as soon as the the analysis is completed and no later than five years after the publication of the trial.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: A fully de-identified data set of the complete patient-level data will be available for sharing purposes as soon as the data analysis is completed and no later than five years after the publication of the trial.
Access Criteria: On request to any interested professional